CLINICAL TRIAL: NCT04416230
Title: The Effects of Massage on Pain After Pediatric Cardiothoracic Surgery
Brief Title: Post-Op Massage in Infants With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Tondi Harrison, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB11-00662
Record Dates: First submitted 2020-05-22; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Congenital Heart Disease
Keywords: congenital heart disease; massage; pediatric pain
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Massage

STUDY DESIGN:
Intervention Model Description: The intervention consisted of a massage given by a licensed massage therapist on each of seven consecutive days beginning on the day of surgery (Day 1). The massage included 30 minutes of Swedish massage on the infant's accessible upper extremities, lower extremities, head, face, and back. Standard precautions were used, including proper hand hygiene and the use of gloves when needed for infection control.
  Infants randomized to the comparison group received a 30 minute quiet time (QT) period during which non-essential caregiving tasks were restricted. During QT, clinicians were asked to avoid direct clinical caregiving activities, i.e. activities requiring physical contact with the infant.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Research assistants scoring participant pain were blinded to group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage (Experimental): Infants randomized to the massage intervention received a 30 minute massage daily for the 7 day study.
  Interventions: Behavioral: massage
- Quiet Time (Active Comparator): Infants randomized to the Quiet Time intervention experienced a 30 minute time during which non-essential clinical caregiving tasks were restricted.
  Interventions: Behavioral: quiet time

INTERVENTIONS:
Behavioral: massage — The massage included 30 minutes of gentle friction, kneading, stroking, and passive touch on the infant's accessible upper extremities, lower extremities, head, face, and back.
  Arms: Massage
Behavioral: quiet time — During quiet time, the infant received a 30 minute quiet time (QT) period during which non-essential caregiving tasks were restricted. During QT, clinicians were asked to avoid direct clinical caregiving activities, i.e. activities requiring physical contact with the infant.
  Arms: Quiet Time

SUMMARY:
The primary aims of the proposed study are to pilot test the effectiveness of daily massage on pain and clinical outcomes in infants who have undergone cardiothoracic surgery. The secondary aim is to explore relationships among massage, pain scores, and other variables potentially affecting pain scores, including parental anxiety, severity of cardiac defect, and severity of pain.

Specific Aim 1: To compare effects of massage on infant pain and clinical outcomes between two groups over time: infants receiving post-operative massage seven days post-operatively and infants receiving a comparable time of restricted non-essential caregiving seven days post-operatively.

Specific Aim 2: To compare pain scores and physiologic responses before and after intervention in two groups: infants receiving post-operative massage and infants receiving a comparable time of restricted non-essential caregiving.

Specific Aim 3: To examine potential moderators of pain response in the massage intervention group before and after receiving massage.

DETAILED DESCRIPTION:
We used a two-group randomized clinical trial design with a sample of 60 infants with complex congenital heart disease (CCHD) between 1 day and 12 months of age following their first cardiothoracic surgery. Both groups received standard post-operative care. In addition, Group 1 received a daily 30-minute restricted non-essential direct caregiving time (Quiet Time), and Group 2 received a daily 30-minute massage. Interventions continued for seven consecutive days. Pain was measured 6 times daily using the Face, Legs, Activity, Cry, Consolability Pain Assessment Tool (FLACC). Average daily doses of analgesics were recorded. Heart rates (HR), respiratory rates (RR), and oxygen saturations (SpO2) were recorded continuously. Daily averages and pre- and post- intervention FLACC scores and physiologic responses were analyzed using descriptive statistics, generalized linear mixed models (GLMM) for repeated measures, latent growth models, and/or regression discontinuity analysis. Fentanyl-equivalent narcotic values were used as a time-varying covariate.

ELIGIBILITY:
Inclusion Criteria:

* Infants born with complex congenital heart disease requiring surgical intervention
* less than 12 months old
* undergoing first surgical procedure

Exclusion Criteria:

* on paralytics post-operatively
* cardiorespiratory instability
* on-going cardiac pacing

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2013-08-03 (Actual); Study Completion 2014-05-30 (Actual)

PRIMARY OUTCOMES:
Post-operative pain score | Daily average for 7 days
  FLACC score: behavioral observation of face, legs, activity, cry, consolability
Change in post-operative pain score with intervention | Daily for 7 days
  FLACC score: behavioral observation of face, legs, activity, cry, consolability
Heart rate | Daily average for 7 days
  heart rate in beats per minute
Respiratory rate | Daily average for 7 days
  respiratory rate in breaths per minute
Oxygen saturation | Daily average for 7 days
  oxygen saturation percentage
Change in heart rate with intervention | Daily for 7 days
  heart rate in beats per minute
Change in respiratory rate with intervention | Daily for 7 days
  respiratory rate in beats per minute
Change in oxygen saturation with intervention | Daily for 7 days
  oxygen saturation percentage

CONTACTS AND LOCATIONS:
Overall Officials: Tondi M Harrison, PhD, RN, Principal Investigator — The Ohio State University and Nationwide Children's Hospital

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Background] Blakely WP, Page GG. Pathophysiology of pain in critically ill patients. Crit Care Nurs Clin North Am. 2001 Jun;13(2):167-79. No abstract available. PMID 11866400
- [Background] Craig KD, Whitfield MF, Grunau RVE, Linton J, Hadjistavropoulos HD. Pain in the preterm neonate: behavioural and physiological indices. Pain. 1993 Mar;52(3):287-299. doi: 10.1016/0304-3959(93)90162-I. PMID 8460047
- [Background] Messerer B, Gutmann A, Weinberg A, Sandner-Kiesling A. Implementation of a standardized pain management in a pediatric surgery unit. Pediatr Surg Int. 2010 Sep;26(9):879-89. doi: 10.1007/s00383-010-2642-1. Epub 2010 Jul 13. PMID 20625751
- [Background] Kulkarni A, Kaushik JS, Gupta P, Sharma H, Agrawal RK. Massage and touch therapy in neonates: the current evidence. Indian Pediatr. 2010 Sep;47(9):771-6. PMID 21048258
- [Background] Mitchinson AR, Kim HM, Rosenberg JM, Geisser M, Kirsh M, Cikrit D, Hinshaw DB. Acute postoperative pain management using massage as an adjuvant therapy: a randomized trial. Arch Surg. 2007 Dec;142(12):1158-67; discussion 1167. doi: 10.1001/archsurg.142.12.1158. PMID 18086982
- [Background] Piotrowski MM, Paterson C, Mitchinson A, Kim HM, Kirsh M, Hinshaw DB. Massage as adjuvant therapy in the management of acute postoperative pain: a preliminary study in men. J Am Coll Surg. 2003 Dec;197(6):1037-46. doi: 10.1016/j.jamcollsurg.2003.07.020. PMID 14644293
- [Background] Nerbass FB, Feltrim MI, Souza SA, Ykeda DS, Lorenzi-Filho G. Effects of massage therapy on sleep quality after coronary artery bypass graft surgery. Clinics (Sao Paulo). 2010;65(11):1105-10. doi: 10.1590/s1807-59322010001100008. PMID 21243280
- [Background] Bauer BA, Cutshall SM, Wentworth LJ, Engen D, Messner PK, Wood CM, Brekke KM, Kelly RF, Sundt TM 3rd. Effect of massage therapy on pain, anxiety, and tension after cardiac surgery: a randomized study. Complement Ther Clin Pract. 2010 May;16(2):70-5. doi: 10.1016/j.ctcp.2009.06.012. Epub 2009 Jul 14. PMID 20347836
- [Background] Albert NM, Gillinov AM, Lytle BW, Feng J, Cwynar R, Blackstone EH. A randomized trial of massage therapy after heart surgery. Heart Lung. 2009 Nov-Dec;38(6):480-90. doi: 10.1016/j.hrtlng.2009.03.001. Epub 2009 Jun 28. PMID 19944872
- [Background] Hernandez-Reif M, Field T, Largie S, Hart S, Redzepi M, Nierenberg B, Peck TM. Childrens' distress during burn treatment is reduced by massage therapy. J Burn Care Rehabil. 2001 Mar-Apr;22(2):191-5; discussion 190. doi: 10.1097/00004630-200103000-00021. PMID 11302609
- [Background] Field T, Hernandez-Reif M, Seligman S, Krasnegor J, Sunshine W, Rivas-Chacon R, Schanberg S, Kuhn C. Juvenile rheumatoid arthritis: benefits from massage therapy. J Pediatr Psychol. 1997 Oct;22(5):607-17. doi: 10.1093/jpepsy/22.5.607. PMID 9383925
- [Background] Benarroch EE. Pain-autonomic interactions. Neurol Sci. 2006 May;27 Suppl 2:S130-3. doi: 10.1007/s10072-006-0587-x. PMID 16688616
- [Background] Kirchner A, Birklein F, Stefan H, Handwerker HO. Left vagus nerve stimulation suppresses experimentally induced pain. Neurology. 2000 Oct 24;55(8):1167-71. doi: 10.1212/wnl.55.8.1167. PMID 11071495
- [Background] Kirchner A, Stefan H, Bastian K, Birklein F. Vagus nerve stimulation suppresses pain but has limited effects on neurogenic inflammation in humans. Eur J Pain. 2006 Jul;10(5):449-55. doi: 10.1016/j.ejpain.2005.06.005. Epub 2005 Aug 24. PMID 16125425
- [Background] Diego MA, Field T, Hernandez-Reif M. Vagal activity, gastric motility, and weight gain in massaged preterm neonates. J Pediatr. 2005 Jul;147(1):50-5. doi: 10.1016/j.jpeds.2005.02.023. PMID 16027695
- [Background] McCain GC, Ludington-Hoe SM, Swinth JY, Hadeed AJ. Heart rate variability responses of a preterm infant to kangaroo care. J Obstet Gynecol Neonatal Nurs. 2005 Nov-Dec;34(6):689-94. doi: 10.1177/0884217505281857. PMID 16282226
- [Background] Feldman R, Eidelman AI. Skin-to-skin contact (Kangaroo Care) accelerates autonomic and neurobehavioural maturation in preterm infants. Dev Med Child Neurol. 2003 Apr;45(4):274-81. doi: 10.1017/s0012162203000525. PMID 12647930
- [Background] Weissman A, Aranovitch M, Blazer S, Zimmer EZ. Heel-lancing in newborns: behavioral and spectral analysis assessment of pain control methods. Pediatrics. 2009 Nov;124(5):e921-6. doi: 10.1542/peds.2009-0598. Epub 2009 Oct 19. PMID 19841119
- [Background] Oberlander TF, Grunau RE, Fitzgerald C, Whitfield MF. Does parenchymal brain injury affect biobehavioral pain responses in very low birth weight infants at 32 weeks' postconceptional age? Pediatrics. 2002 Sep;110(3):570-6. doi: 10.1542/peds.110.3.570. PMID 12205262
- [Background] Faye PM, De Jonckheere J, Logier R, Kuissi E, Jeanne M, Rakza T, Storme L. Newborn infant pain assessment using heart rate variability analysis. Clin J Pain. 2010 Nov-Dec;26(9):777-82. doi: 10.1097/ajp.0b013e3181ed1058. PMID 20973153
- [Background] Logier R, Jeanne M, Tavernier B, De Jonckheere J. Pain/analgesia evaluation using heart rate variability analysis. Conf Proc IEEE Eng Med Biol Soc. 2006;2006:4303-6. doi: 10.1109/IEMBS.2006.260494. PMID 17946620
- [Background] Anand KJ, Aranda JV, Berde CB, Buckman S, Capparelli EV, Carlo W, Hummel P, Johnston CC, Lantos J, Tutag-Lehr V, Lynn AM, Maxwell LG, Oberlander TF, Raju TN, Soriano SG, Taddio A, Walco GA. Summary proceedings from the neonatal pain-control group. Pediatrics. 2006 Mar;117(3 Pt 2):S9-S22. doi: 10.1542/peds.2005-0620C. PMID 16777824
- [Background] Stapelkamp C, Carter B, Gordon J, Watts C. Assessment of acute pain in children: development of evidence-based guidelines. Int J Evid Based Healthc. 2011 Mar;9(1):39-50. doi: 10.1111/j.1744-1609.2010.00199.x. PMID 21332662
- [Background] Granot M, Ferber SG. The roles of pain catastrophizing and anxiety in the prediction of postoperative pain intensity: a prospective study. Clin J Pain. 2005 Sep-Oct;21(5):439-45. doi: 10.1097/01.ajp.0000135236.12705.2d. PMID 16093750
- [Background] Kalkman JC, Visser K, Moen J, Bonsel JG, Grobbee ED, Moons MKG. Preoperative prediction of severe postoperative pain. Pain. 2003 Oct;105(3):415-423. doi: 10.1016/S0304-3959(03)00252-5. PMID 14527702
- [Background] Bringuier S, Dadure C, Raux O, Dubois A, Picot MC, Capdevila X. The perioperative validity of the visual analog anxiety scale in children: a discriminant and useful instrument in routine clinical practice to optimize postoperative pain management. Anesth Analg. 2009 Sep;109(3):737-44. doi: 10.1213/ane.0b013e3181af00e4. PMID 19690240
- [Background] Franck LS, Ridout D, Howard R, Peters J, Honour JW. A comparison of pain measures in newborn infants after cardiac surgery. Pain. 2011 Aug;152(8):1758-1765. doi: 10.1016/j.pain.2011.03.017. Epub 2011 Apr 21. PMID 21514052
- [Background] Smith MC, Stallings MA, Mariner S, Burrall M. Benefits of massage therapy for hospitalized patients: a descriptive and qualitative evaluation. Altern Ther Health Med. 1999 Jul;5(4):64-71. PMID 10394676
- [Background] Diego MA, Field T, Hernandez-Reif M, Deeds O, Ascencio A, Begert G. Preterm infant massage elicits consistent increases in vagal activity and gastric motility that are associated with greater weight gain. Acta Paediatr. 2007 Nov;96(11):1588-91. doi: 10.1111/j.1651-2227.2007.00476.x. Epub 2007 Sep 21. PMID 17888059
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Voepel-Lewis T, Merkel S, Tait AR, Trzcinka A, Malviya S. The reliability and validity of the Face, Legs, Activity, Cry, Consolability observational tool as a measure of pain in children with cognitive impairment. Anesth Analg. 2002 Nov;95(5):1224-9, table of contents. doi: 10.1097/00000539-200211000-00020. PMID 12401598
- [Background] 32. Wong DL, Hockenberry-Eaton M, Wilson D, et al. Wong's essentials of pediatric nursing (6th ed.). St. Louis: Mosby; 2001.
- [Background] Jensen MP, Karoly P, O'Riordan EF, Bland F Jr, Burns RS. The subjective experience of acute pain. An assessment of the utility of 10 indices. Clin J Pain. 1989 Jun;5(2):153-9. doi: 10.1097/00002508-198906000-00005. PMID 2520397
- [Background] 34. Spielberger CD. Conceptual and methodological issues in anxiety research. In C. D. Spielberger (Ed.), Anxiety: current trends in theory and research (pp. 481-492). New York: Academic Press; 1972.
- [Background] Page MG, Fuss S, Martin AL, Escobar EM, Katz J. Development and preliminary validation of the Child Pain Anxiety Symptoms Scale in a community sample. J Pediatr Psychol. 2010 Nov;35(10):1071-82. doi: 10.1093/jpepsy/jsq034. Epub 2010 Apr 29. PMID 20430838
- [Background] Page GM, Campbell F, Isaac L, Stinson J, Martin-Pichora AL, Katz J. Reliability and validity of the Child Pain Anxiety Symptoms Scale (CPASS) in a clinical sample of children and adolescents with acute postsurgical pain. Pain. 2011 Sep;152(9):1958-1965. doi: 10.1016/j.pain.2011.02.053. Epub 2011 Apr 12. PMID 21489692
- [Background] Jenkins KJ, Gauvreau K, Newburger JW, Spray TL, Moller JH, Iezzoni LI. Consensus-based method for risk adjustment for surgery for congenital heart disease. J Thorac Cardiovasc Surg. 2002 Jan;123(1):110-8. doi: 10.1067/mtc.2002.119064. PMID 11782764
- [Derived] Harrison TM, Brown R, Duffey T, Frey C, Bailey J, Nist MD, Renner L, Fitch J. Effects of Massage on Postoperative Pain in Infants With Complex Congenital Heart Disease. Nurs Res. 2020 Sep/Oct;69(5S Suppl 1):S36-S46. doi: 10.1097/NNR.0000000000000459. PMID 32858717